CLINICAL TRIAL: NCT03119350
Title: Mitochondrial Energy Metabolism in Obese Women Undergoing Concurrent Physical Training
Brief Title: Mitochondrial Energy Metabolism in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Julio Sergio Marchini, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Process HCRP: 1.387.040/2016
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Metabolism Disorder; Mitochondrial Alteration; Physical Activity; Obesity
MeSH Terms: conditions — Metabolic Diseases; Motor Activity; Obesity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Training (Other): There was concurrent physical training intervention: strength and aerobic exercises in the same session.
  Duration: 2 weeks of adaptation and learning to exercise, 8 weeks of physical training.
  Frequency: 3 times per week Duration: 55 minutes each session. Intensity: 75 to 90% of maximum heart rate.
  Interventions: Other: Physical Training

INTERVENTIONS:
Other: Physical Training — Intervention with concurrent physical training: strength and aerobic exercises in the same session.
  Duration: 2 weeks of adaptation to physical exercise, 8 weeks of training. Frequency: 3 times a week. Time: 55 minutes each session. Intensity: 75 to 90% of maximum heart rate.

SUMMARY:
Considering that the failure of the treatment of obesity is justified by the multifactorial pathophysiology of this morbidity, the present project has the following hypotheses:

1. The occurrence of obesity is due to the derange,ent of mitochondrial energy metabolism ;
2. The unbalance is therapeutically modified through physical training ;
3. Obesity courses with the break-down in energy metabolism mitochondrial disease associated with systemic inflammatory characteristics that can be corrected through a combined long-term physical training program.

This study have as objective : to analyse changes in mitochondrial function, inflammatory profile, oxidative stress and energy metabolism caused by concurrent physical training in obese women.

DETAILED DESCRIPTION:
Specific objectives:

Body composition by deuterium oxide; Metabolic rate of resting and oxidation of substrates by indirect calorimetry; Proinflammatory cytokines Anti-inflammatory cytokines Oxidative Stress: Malondialdehyde, Superoxide Dismutase, Glutathione-Peroxidase; Fatty acids: ceramide and palmitate; Mitochondrial respiration and citrate synthase enzyme; Quantify and qualify: mitochondrial number, endoplasmic reticulum structure, adipose cell size; Gene expression, quantify by microscopy and analyze the protein by western blot.

The study began with 20 women, however, there was withdrawal of 6, ending with 14 women.

ELIGIBILITY:
Inclusion Criteria:

* This study included women with obesity (BMI of 30 to 40 kg / m²), sedentary, with no associated comorbidity, convenience sample

Exclusion Criteria:

* Women who have undergone bariatric surgery, menopause, cancer or any metabolic disease, smokers, alcoholics, who are in use of drugs that act directly on the metabolism and that have medical impediment to the practice of physical exercise.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Changes Body weight | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Body weight was measured by digital balance before and after the intervention
Changes Body composition | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  The change in body composition through deuterium oxide was evaluated.
Changes White adipose tissue biopsy | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  A subcutaneous tissue sample was collected for analysis of: mitochondrial respiration, citrate synthase enzyme, gene expression (UCP1, 2 and 3).
Changes Indirect calorimetry | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  With a gas analyzer (indirect calorimeter), we evaluated the metabolic rate and rest (REE) and oxidation of substrates (Lipids and carbohydrates).
Changes in fatty acids | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Collected in lithium heparin tubes, they were centrifuged.
Changes oxidative stress | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Collected in lithium heparin tubes, they were centrifuged.
Changes inflammatory cytokines | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Collected in lithium heparin tubes, they were centrifuged.
Changes in total cholesterol | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Collected in lithium heparin tubes, they were centrifuged.
Changes Physical Performance | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Based on the Shuttle Walking Test adaptation.
Changes in Determination of Lactate | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Blood samples were collected by manual puncture of the earlobe in previously calibrated and heparinized capillary tubes, stored in eppendorf with sodium fluoride. Analyzed by electrochemical lactate analyser.
Changes Food intake | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Food registry of 3 days, the quantification of the daily intake of nutrients will still be made using software.
Changes Nitrogen Balance | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  Through the collection of urine of 24 hours the dosage of urinary nitrogen will be made by the chemiluminescence method for determination of protein nitrogen.
Changes Telomere length | Two times: (1) First day and (2) 10 weeks after adaptation and intervention
  peripheral blood in ethylenediaminetetraacetic acid tubes and genomic DNA was automatically extracted from Peripheral Blood Mononuclear Cell. The relative quantification of Telomere length was determined using the telomere to single copy gene ratio by Quantitative Polymerase Chain Reaction (qPCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Camila Fernanda Cunha Brandão, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BROWN, L.E.; WEIR, J.P.; ASEP procedures recommendation i: accurate assessment of muscular strength and power, Journal of Exercise Physiology, v. 4, n. 3, p. 1-21, 2001.
- [Background] Burgomaster KA, Howarth KR, Phillips SM, Rakobowchuk M, Macdonald MJ, McGee SL, Gibala MJ. Similar metabolic adaptations during exercise after low volume sprint interval and traditional endurance training in humans. J Physiol. 2008 Jan 1;586(1):151-60. doi: 10.1113/jphysiol.2007.142109. Epub 2007 Nov 8. PMID 17991697
- [Background] Chomczynski P, Sacchi N. Single-step method of RNA isolation by acid guanidinium thiocyanate-phenol-chloroform extraction. Anal Biochem. 1987 Apr;162(1):156-9. doi: 10.1006/abio.1987.9999. PMID 2440339
- [Background] Colégio Americano de Medicina Esportiva, CAME. Guia para Teste de Esforço e Prescrição de Exercício. 3º Edição, Medsi, Rio de janeiro, RJ, p.25, 1987.
- [Background] Crump C, Sundquist J, Winkleby MA, Sundquist K. Interactive effects of obesity and physical fitness on risk of ischemic heart disease. Int J Obes (Lond). 2017 Feb;41(2):255-261. doi: 10.1038/ijo.2016.209. Epub 2016 Nov 21. PMID 27867205
- [Background] Curtis JM, Grimsrud PA, Wright WS, Xu X, Foncea RE, Graham DW, Brestoff JR, Wiczer BM, Ilkayeva O, Cianflone K, Muoio DE, Arriaga EA, Bernlohr DA. Downregulation of adipose glutathione S-transferase A4 leads to increased protein carbonylation, oxidative stress, and mitochondrial dysfunction. Diabetes. 2010 May;59(5):1132-42. doi: 10.2337/db09-1105. Epub 2010 Feb 11. PMID 20150287
- [Background] Daussin FN, Zoll J, Dufour SP, Ponsot E, Lonsdorfer-Wolf E, Doutreleau S, Mettauer B, Piquard F, Geny B, Richard R. Effect of interval versus continuous training on cardiorespiratory and mitochondrial functions: relationship to aerobic performance improvements in sedentary subjects. Am J Physiol Regul Integr Comp Physiol. 2008 Jul;295(1):R264-72. doi: 10.1152/ajpregu.00875.2007. Epub 2008 Apr 16. PMID 18417645
- [Background] EIGENTLER, A.; DRAXL, A.; et al. Laboratory Protocol: Citrate synthase a mitochondrial marker enzyme. Mitochondrial Physiology Network, v. 17.04, n. 3, p. 1-11, 2015.
- [Background] Fernstrom M, Bakkman L, Loogna P, Rooyackers O, Svensson M, Jakobsson T, Brandt L, Lagerros YT. Improved Muscle Mitochondrial Capacity Following Gastric Bypass Surgery in Obese Subjects. Obes Surg. 2016 Jul;26(7):1391-7. doi: 10.1007/s11695-015-1932-z. PMID 26471784
- [Background] Ferreira FC, Bertucci DR, Barbosa MR, Nunes JE, Botero JP, Rodrigues MF, Shiguemoto GE, Santoro V, Verzola AC, Nonaka RO, Verzola RM, Baldissera V, Perez SE. Circuit resistance training in women with normal weight obesity syndrome: body composition, cardiometabolic and echocardiographic parameters, and cardiovascular and skeletal muscle fitness. J Sports Med Phys Fitness. 2017 Jul-Aug;57(7-8):1033-1044. doi: 10.23736/S0022-4707.16.06391-X. Epub 2016 Jul 6. PMID 27385544
- [Background] FETT, C.A.; FETT, W.C.R.; MARCHINI, J.S. Fitness Level of Overweight/Obese Women After 08 Weeks of Aerobic or Mixed Metabolism Exercises. Revista Brasileira de Cineantropometria & Desempenho Humano, v. 11, p. 261-266, 2009.
- [Background] Foster C. Monitoring training in athletes with reference to overtraining syndrome. Med Sci Sports Exerc. 1998 Jul;30(7):1164-8. doi: 10.1097/00005768-199807000-00023. PMID 9662690
- [Background] Frayn KN. Calculation of substrate oxidation rates in vivo from gaseous exchange. J Appl Physiol Respir Environ Exerc Physiol. 1983 Aug;55(2):628-34. doi: 10.1152/jappl.1983.55.2.628. PMID 6618956
- [Background] Grimble GK, West MF, Acuti AB, Rees RG, Hunjan MK, Webster JD, Frost PG, Silk DB. Assessment of an automated chemiluminescence nitrogen analyzer for routine use in clinical nutrition. JPEN J Parenter Enteral Nutr. 1988 Jan-Feb;12(1):100-6. doi: 10.1177/0148607188012001100. PMID 3125351
- [Background] Heilbronn LK, Gan SK, Turner N, Campbell LV, Chisholm DJ. Markers of mitochondrial biogenesis and metabolism are lower in overweight and obese insulin-resistant subjects. J Clin Endocrinol Metab. 2007 Apr;92(4):1467-73. doi: 10.1210/jc.2006-2210. Epub 2007 Jan 23. PMID 17244782
- [Background] Koh EH, Park JY, Park HS, Jeon MJ, Ryu JW, Kim M, Kim SY, Kim MS, Kim SW, Park IS, Youn JH, Lee KU. Essential role of mitochondrial function in adiponectin synthesis in adipocytes. Diabetes. 2007 Dec;56(12):2973-81. doi: 10.2337/db07-0510. Epub 2007 Sep 7. PMID 17827403
- [Background] Kong Z, Sun S, Liu M, Shi Q. Short-Term High-Intensity Interval Training on Body Composition and Blood Glucose in Overweight and Obese Young Women. J Diabetes Res. 2016;2016:4073618. doi: 10.1155/2016/4073618. Epub 2016 Sep 28. PMID 27774458
- [Background] Kraunsoe R, Boushel R, Hansen CN, Schjerling P, Qvortrup K, Stockel M, Mikines KJ, Dela F. Mitochondrial respiration in subcutaneous and visceral adipose tissue from patients with morbid obesity. J Physiol. 2010 Jun 15;588(Pt 12):2023-32. doi: 10.1113/jphysiol.2009.184754. Epub 2010 Apr 26. PMID 20421291
- [Background] Lepage G, Roy CC. Improved recovery of fatty acid through direct transesterification without prior extraction or purification. J Lipid Res. 1984 Dec 1;25(12):1391-6. PMID 6530596
- [Background] Medbo JI, Mamen A, Holt Olsen O, Evertsen F. Examination of four different instruments for measuring blood lactate concentration. Scand J Clin Lab Invest. 2000 Aug;60(5):367-80. doi: 10.1080/003655100750019279. PMID 11003256
- [Background] Perry CG, Lally J, Holloway GP, Heigenhauser GJ, Bonen A, Spriet LL. Repeated transient mRNA bursts precede increases in transcriptional and mitochondrial proteins during training in human skeletal muscle. J Physiol. 2010 Dec 1;588(Pt 23):4795-810. doi: 10.1113/jphysiol.2010.199448. Epub 2010 Oct 4. PMID 20921196
- [Background] Pfrimer K, Moriguti JC, Lima NK, Marchini JS, Ferriolli E. Bioelectrical impedance with different equations versus deuterium oxide dilution method for the inference of body composition in healthy older persons. J Nutr Health Aging. 2012 Feb;16(2):124-7. doi: 10.1007/s12603-011-0137-y. PMID 22323345
- [Background] POLLOCK, M.L.; WILMORE, J.H.; FOX III, S.M. Exercícios na Saúde e na Doença - Avaliação e prescrição para prevenção e reabilitação. Rio de Janeiro: 1986.
- [Background] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Background] Tan S, Wang J, Cao L, Guo Z, Wang Y. Positive effect of exercise training at maximal fat oxidation intensity on body composition and lipid metabolism in overweight middle-aged women. Clin Physiol Funct Imaging. 2016 May;36(3):225-30. doi: 10.1111/cpf.12217. Epub 2014 Nov 19. PMID 27072372
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301
- [Background] Yin X, Lanza IR, Swain JM, Sarr MG, Nair KS, Jensen MD. Adipocyte mitochondrial function is reduced in human obesity independent of fat cell size. J Clin Endocrinol Metab. 2014 Feb;99(2):E209-16. doi: 10.1210/jc.2013-3042. Epub 2013 Nov 25. PMID 24276464
- [Derived] Brandao CFC, Nonino CB, de Carvalho FG, Nicoletti CF, Noronha NY, San Martin R, de Freitas EC, Junqueira-Franco MVM, Marchini JS. The effects of short-term combined exercise training on telomere length in obese women: a prospective, interventional study. Sports Med Open. 2020 Jan 16;6(1):5. doi: 10.1186/s40798-020-0235-7. PMID 31950310